CLINICAL TRIAL: NCT04618978
Title: Periodic Leg Movement's Diagnosis in Spinal Cord Injury: Actigraphy as an Alternative for Polysomnography?
Brief Title: Periodic Leg Movements' Diagnosis in Spinal Cord Injury: Actigraphy as an Alternative for Polysomnography?
Acronym: ACTI-MPJ-BM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP200140
Record Dates: First submitted 2020-10-23; First posted 2020-11-06 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-01

CONDITIONS: Spinal Cord Injuries; Periodic Limb Movement Disorder
Keywords: spinal cord injury; multiple sclerosis; periodic leg movements; spasticity; periodic limb movement disorder
MeSH Terms: conditions — Spinal Cord Injuries; Nocturnal Myoclonus Syndrome; Multiple Sclerosis; Muscle Spasticity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PSG and actigraphy device evaluations (Other): All patients will be evaluated and diagnosed according to the records by Gold standard for PLMs diagnosis and also by the actigraphy devices recording.
  Interventions: Procedure: PSG and actigraphy recording

INTERVENTIONS:
Procedure: PSG and actigraphy recording — Gold standard: electromyographic recording of tibialis anterior muscle during full night polysomnography (PSG).
  The new generation actigraphs devices Actiwatch will be combined to PSG as a screening tool: MotionWatch will be placed on the dorsum of feet to record).

SUMMARY:
Periodic Limb Movements during Sleep (PLMs) are episodes of repetitive, stereotypical, hallux or foot movements. They could induce sleep disturbance, fatigue, daytime sleepiness and impaired quality of life but also increased cardiovascular risk by rising heart rate and blood pressure at night. Gold standard for PLMs diagnosis is based on electromyographic recording of tibialis anterior muscle during full night polysomnography (PSG).

PLMs prevalence is higher in patients with spinal cord injury (SCI) possibly due to a loss of encephalic inhibition on a spinal motion generator. In these patients, PLMs can also be wrongly considered as spasms sometimes leading to the unjustified implantation of an intrathecal Lioresal pump.

In the general population, drug treatments for PLMs, particularly dopamine agonists, limit the impact of these abnormal movements on sleep fragmentation, daytime alertness and quality of life. Underdiagnosed PLMs in SCI patients can lead to exacerbate cognitive, mood and painful disorders due to the close interaction between sleep disorders and neurocognitive, psychological and painful manifestations.

PLMs appropriate diagnosis appeared mandatory in those patients but accessibility and delayed availability remain challenging. In addition, sleep laboratories are often unable to accommodate with SCI patients.

In this context, actigraphy, an easy-to-use, cheaper and easily renewable diagnostic tool would be interesting. In the general population, sensitivity to diagnose PLMs was between 0.79 and 1 and specificity between 0.6 and 0.83. Due to lower limbs impairment, increased specificity is expected SCI patients (decrease voluntary activity).

The new generation of actigraph (MotionWatchR) could have better characteristics thanks to the development of a specific software which integrate both lower limbs in the same analysis.

As primary objective, this prospective monocentric study aims to evaluate the performances of lower limbs actigraphy for PLMs diagnosis versus gold standard.

DETAILED DESCRIPTION:
As secondary objectives, the study aims to:

* Estimate positive and negative predictive values;
* Identify the diagnostic threshold of PLMs index with actigraphy;
* Study concordance between actigraphy and polysomnography to detect lower limbs movements;
* Evaluate reproducibility between 2 readers and with the new PLMs software;
* Study actigraphy reproducibility for this indication over 3 consecutive nights in the same patients (ancillary study);
* Compare diagnostic performance according to SCI completeness (AIS-A vs AIS-B, C, D) and underlying pathology (MS, SCI);
* Compare installation and interpretation times between actigraphy and PSG.

PLMs appropriate diagnosis appeared mandatory in SCI patients however the accessibility and the delay of availability remain challenging for severe SCI complications in care management.

The study team hypothesize that actigraphy could be able to diagnose PLMs with sufficient reliability (AUC (area under the curve) around 80%) compared to the gold standard (polysomnography) in patients with spinal cord injuries.

Intervention: During a scheduled night recording (polysomnography) 3 actigraphs will be added (1 on the wrist, and 1 on each foot).

Equipment: MotionWatch8®, CamNtech® (marking CE Class 1 device; accord FDA (K132764)).

Methods:

All consecutive eligible patients followed in our tertiary care center (for whom a full night polysomnography is already scheduled) will be informed of the study and proposed to participate.

After signing the informed consent form, all subjects will undergo a full-night examinations: polysomnography (already scheduled in usual care) and actigraphy (addition of 3 devices):

* 1 classic actigraph on the wrist to detect light and identify inactivity periods compatible with sleep.
* 2 new generation Actiwatch actigraphs (MotionWatch) placed on the feet. Polysomnography will incorporate tibialis anterior EMG recording and will be scored by one sleep specialist following American Academy of Sleep Medicine (AASM) scoring criteria.

Actigraphy analysis will be provided by:

* An automated software specially developed for this indication (PLMsanalysis software, camNtechR).
* A nurse reading unaware of both software's and PSG results.
* A second reading will be provided by a second nurse, also unaware of the result of the polysomnography.

Actigraphy results will not be communicated to patients or physicians and therefore will not affect patient management.

At the end of the evaluation period, each patient will be offered, if needed, treatment and follow-up in the sleep unit as in usual care.

A study of actigraphy reproducibility will be carried out in a sample of 33 subjects. This study will take place over three consecutive nights during an already scheduled hospitalization (no additional hospitalization night for patients).

Statistical analysis: as described in Outcome Measures.

ELIGIBILITY:
Inclusion Criteria:

* Patient With Spinal Cord Injury from traumatic or medical aetiology (including patient with multiple sclerosis);
* Motor testing stability for at least 6 months prior to inclusion;
* Patients with complete or incomplete SCI (AIS-A, B, C, D and E);
* Neurological level between C4 and L1;
* Aged >18 years;
* Patients with already scheduled full night polysomnography (PSG);
* Affiliated to social security system;
* Absence of medical intercurrent event.

Exclusion Criteria:

Specific criteria:

* History of lower limbs amputation ;
* Cutaneous lesion compromising actigraphy positioning
* Presence of spinal cord stimulation equipment, Brindley electrodes, history of spinal cord surgery.

No-specific criteria:

* Patient refusal;
* Participation in another interventional study involving human participants
* Unable to sign informed consent form;
* Emergency condition;
* Legal protection (i.e. incompetence to provide consent, guardianship, curator or incarceration);
* No affiliation to a social security system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2024-07-04 (Actual); Study Completion 2025-01-17 (Actual)

PRIMARY OUTCOMES:
The Receiver Operating Characteristic (ROC) analysis | Through study completion, an average of 3 years
  Area under ROC curve of the actimeter (indices of periodic movement of legs, defined by the ratio between the number of periodic movement of low limbs during sleeping time and estimated sleeping duration in hour), compared with polysomnography to have diagnosis of periodic movement of legs during sleeping (period of sleeping defined by absence of light and movement of up limb of the more mobile with actimeter).

SECONDARY OUTCOMES:
Predictive values estimation | Through study completion, an average of 3 years
  Sensitivity, specificity, positive and negative predictive values and likelihood ratio of actigraphy compared to polysomnography to diagnose PLMs
Threshold of PLMs Index | up to 24 hours
  The periodic limb movement index (PLMI), which corresponds to the number of periodic limb movements per hour.
  The actigraphy will be used to determinate diagnostic threshold of PLMs Index.
Lower limb nocturnal movements evaluation | up to 24 hours
  Number of lower limb nocturnal movements per recording hour
PLMs diagnosis based on the actigraphy | Through study completion, an average of 3 years
  PLMs diagnosis (yes / no) based on the actigraphy results
Kappa coefficient | Through study completion, an average of 3 years
  Kappa coefficient between PLMs diagnoses (yes / no) made by 2 different nurses and between 1 nurse and the automated analysis software
Actigraphy diagnostic performance | Through study completion, an average of 3 years
  Actigraphy diagnostic performance according to:
  * the underlying pathology (MS or not)
  * and lesion completeness (AIS-A vs AIS-B,C, D)
  AIS: American Spinal Injury Association (ASIA) Impairment Scale;
  MS: multiple sclerosis.
Installation time | Through study completion, an average of 3 years
  Installation time between actigraphy and PSG
Interpretation time | Through study completion, an average of 3 years
  Time of interpretation between actigraphy and PSG

CONTACTS AND LOCATIONS:
Overall Officials: Marie Christine BLANDIN, Principal Investigator — Physiologie, explorations fonctionnelles - Unité des pathologies du sommeil, Hôpital Raymond Poincaré, APHP; Antoine LEOTARD, MD, Study Director — Physiologie, explorations fonctionnelles - Unité des pathologies du sommeil, Hôpital Raymond Poincaré, APHP
Locations (1):
- Physiologie, explorations fonctionnelles - Unité des pathologies du sommeil, Hôpital Raymond Poincaré, APHP, Garches, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siddiqui F, Strus J, Ming X, Lee IA, Chokroverty S, Walters AS. Rise of blood pressure with periodic limb movements in sleep and wakefulness. Clin Neurophysiol. 2007 Sep;118(9):1923-30. doi: 10.1016/j.clinph.2007.05.006. Epub 2007 Jun 27. PMID 17588809
- [Background] Proserpio P, Lanza A, Sambusida K, Fratticci L, Frigerio P, Sommariva M, Stagni EG, Redaelli T, De Carli F, Nobili L. Sleep apnea and periodic leg movements in the first year after spinal cord injury. Sleep Med. 2015 Jan;16(1):59-66. doi: 10.1016/j.sleep.2014.07.019. Epub 2014 Oct 7. PMID 25454844
- [Background] Foschi M, Rizzo G, Liguori R, Avoni P, Mancinelli L, Lugaresi A, Ferini-Strambi L. Sleep-related disorders and their relationship with MRI findings in multiple sclerosis. Sleep Med. 2019 Apr;56:90-97. doi: 10.1016/j.sleep.2019.01.010. Epub 2019 Jan 21. PMID 30803830
- [Background] Telles SC, Alves RS, Chadi G. Spinal cord injury as a trigger to develop periodic leg movements during sleep: an evolutionary perspective. Arq Neuropsiquiatr. 2012 Nov;70(11):880-4. doi: 10.1590/s0004-282x2012001100011. PMID 23175202
- [Background] Levy J, Hartley S, Mauruc-Soubirac E, Leotard A, Lofaso F, Quera-Salva MA, Bensmail D. Spasticity or periodic limb movements? Eur J Phys Rehabil Med. 2018 Oct;54(5):698-704. doi: 10.23736/S1973-9087.17.04886-9. Epub 2017 Dec 4. PMID 29205982
- [Background] Allen R. Dopamine and iron in the pathophysiology of restless legs syndrome (RLS). Sleep Med. 2004 Jul;5(4):385-91. doi: 10.1016/j.sleep.2004.01.012. PMID 15222997
- [Background] Guilleminault C, Flagg W. Effect of baclofen on sleep-related periodic leg movements. Ann Neurol. 1984 Mar;15(3):234-9. doi: 10.1002/ana.410150304. PMID 6721446
- [Background] Plante DT. Leg actigraphy to quantify periodic limb movements of sleep: a systematic review and meta-analysis. Sleep Med Rev. 2014 Oct;18(5):425-34. doi: 10.1016/j.smrv.2014.02.004. Epub 2014 Feb 17. PMID 24726711
- [Background] Kobayashi M, Namba K, Ito E, Nishida S, Nakamura M, Ueki Y, Furudate N, Kagimura T, Usui A, Inoue Y. The validity of the PAM-RL device for evaluating periodic limb movements in sleep and an investigation on night-to-night variability of periodic limb movements during sleep in patients with restless legs syndrome or periodic limb movement disorder using this system. Sleep Med. 2014 Jan;15(1):138-43. doi: 10.1016/j.sleep.2013.08.790. Epub 2013 Oct 31. PMID 24269130
- [Background] Ferri R, Fulda S, Manconi M, Hogl B, Ehrmann L, Ferini-Strambi L, Zucconi M. Night-to-night variability of periodic leg movements during sleep in restless legs syndrome and periodic limb movement disorder: comparison between the periodicity index and the PLMS index. Sleep Med. 2013 Mar;14(3):293-6. doi: 10.1016/j.sleep.2012.08.014. Epub 2012 Oct 12. PMID 23068780